CLINICAL TRIAL: NCT02394327
Title: Endoscopic Naso-gallbladder Drainage Versus Gallbladder Stenting Before Elective Cholecystectomy in Patients With Acute Cholecystitis and a High Suspicion of Common Bile Duct Stone; A Prospective Randomized Preliminary Study
Brief Title: Endoscopic Nasogallbladder Drainage Versus Gallbladder Stenting Before Cholecystecomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Yoo Byung Moo, Associate professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AJIRB-MED-MDB-11-318
Record Dates: First submitted 2015-02-18; First posted 2015-03-20 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Cholecystitis, Acute; Common Bile Duct Calculi
MeSH Terms: conditions — Cholecystitis, Acute; Gallstones

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Endoscopic nasogallbladder drainage (Active Comparator): If GB cannulation was achieved and the wire was coiled in the GB, 5 to 7-Fr Pigtail type naso-cholecystic drainage tube (Liguory nasal biliary drainage set; Wilson-Cook Medical, Salem, NC, USA) was placed into the GB
  Interventions: Device: 7-Fr Pigtail type naso-cholecystic drainage tube (Liguory nasal biliary drainage set; Wilson-Cook Medical, Salem, NC, USA)
- Endoscopic gallbladder stenting (Active Comparator): If GB cannulation was achieved and the wire was coiled in the GB, 7-Fr double pigtail plastic stent (Zimmon; Wilson-Cook Medical, Salem, NC, USA) was placed into the GB
  Interventions: Device: 7-Fr double pigtail plastic stent (Zimmon; Wilson-Cook Medical, Salem, NC, USA)

INTERVENTIONS:
Device: 7-Fr Pigtail type naso-cholecystic drainage tube (Liguory nasal biliary drainage set; Wilson-Cook Medical, Salem, NC, USA) — Endoscopic
  Arms: Endoscopic nasogallbladder drainage
Device: 7-Fr double pigtail plastic stent (Zimmon; Wilson-Cook Medical, Salem, NC, USA)
  Arms: Endoscopic gallbladder stenting

SUMMARY:
Early laparoscopic cholecystectomy is the current standard therapy for acute cholecystitis, but temporary decompression of the gallbladder (GB) through percutaneous or endoscopic route can be required to alleviate inflammatory process and reach an appropriate time for elective surgery in patients with high operative risk or marked local inflammation or organ dysfunction. Also preoperative endoscopic retrograde cholangiopancreatography (ERCP) is often needed because common bile duct (CBD) stone is accompanied in patients with acute cholecystitis at reported rate from 7-20%.

Two-steps approach of percutaneous transhepatic GB drainage (PTGBD) followed by ERCP or vice versa has been performed for the treatment of acute cholecystitis with concomitant CBD stone who are not suitable for urgent cholecystectomy. However single-step drainage of CBD and GB through ERCP and endoscopic transpapillary GB drainage (ETGD) using nasocystic tube or plastic stent has alternatively been attempted in patients who have contraindications for PTGBD. In clinical practice, many endoscopists have hesitated to perform ETGD because of its relatively low technical success rate and specific concern about post-ERCP adverse event but it minimizes catheter keeping duration, and provides effective clinical improvement via physiologic route.

Currently there are scarce data on if ETGD using nasocystic tube or plastic stent are comparable in terms of clinical efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* grade II or III acute cholecystitis met Tokyo 13 diagnostic criteria
* a high suspicion of CBD stone based on laboratory and imaging study
* informed consent given.

Exclusion Criteria:

* bilo-pancreatic malignancy or surgically altered enteric anatomy
* subsequent elective surgery is expected to be impossible even after GB decompression based on American Society of Anesthesiologist class

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Techncal success rate | From the time of randomization until the time when the endoscopic procedure is ended, assessed up to 24hours
  This outcome was defined as successful deep GB cannulation and placement of assigned drainage device by randomization, and determined by the operator based on the fluoroscoic images of the procedures.

SECONDARY OUTCOMES:
Clinical success rate | From the date of randomization until the date of clinical improvement (fever, leukocytosis, abdominal pain), assessed up to 72 hours
  This outcome was defined as improvement of three clinical parameters of acute cholecystitis (fever, abdominal pain, leukocytosis) within 72 hours following either type of ETGD procedure, and assessed by the review of patient's mediacal records.
early adverse event | From the date of the randomization until the date of the elective cholecystectomy, assessed up to 2 weeks
  This outcome was defined as any procedure related event occurring between the endoscopic procedure and elective cholecystectomy, and assessed by the patient's medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Byung Moo Yoo, MD, Study Director — Ajou University School of Medicine
Locations (1):
- Ajou University Hospital, Suwon, Gyeonggido, South Korea